CLINICAL TRIAL: NCT03911310
Title: [18F]PSMA-11 PET/CT for Prostate Cancer - Phase 3 Clinical Study
Brief Title: [18F]PSMA-11 PET/CT Phase 3 Clinical Study
Acronym: NGP3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AGO/2018/003
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; biochemical recurrence; 18F-PSMA PET imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial encompasses a double-blind randomized cross-over design whereby each patient will be subjected to a [18F]PSMA-11 scan and a [68Ga]PSMA-11 scan, with an interscan period of four days to maximum three weeks. Half of the patients will be first scanned with [18F]PSMA-11 and subsequently (maximum three weeks later) with [68Ga]PSMA-11. The scan order in the remaining group of patients will be reversed. Randomization of patients to one of these groups will be performed using a block randomization design with block sizes of six.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The assigned scan order will be blind to the recruiting physicians and the nuclear medicine physicians interpreting the images.
  Next to the clinical trial coordinators, also the staff members responsible for the preparation of the individual [18F]PSMA-11 and [68Ga]PSMA-11 dose and the IV injection of this dose are aware of the scan order which means that they are NOT blinded. However, these staff members do not carry out any further study specific handlings.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PET/CT 1: [18F]PSMA-11, PET/CT 2: [68Ga]PSMA-11 (Experimental): Patients in this arm will first receive the experimental radiotracer [18F]PSMA-11 PET/CT followed by the [68Ga]PSMA-11 PET/CT after at least 4 days and maximum 3 weeks.
  Interventions: Diagnostic Test: [18F]PSMA-11; Diagnostic Test: [68Ga]PSMA-11
- PET/CT 1: [68Ga]PSMA-11, PET/CT 2: [18F]PSMA-11 (Active Comparator): Patients in this arm will first receive the experimental radiotracer [68Ga]PSMA-11 PET/CT followed by the [18F]PSMA-11 PET/CT after at least 4 days and maximum 3 weeks.
  Interventions: Diagnostic Test: [18F]PSMA-11; Diagnostic Test: [68Ga]PSMA-11

INTERVENTIONS:
Diagnostic Test: [18F]PSMA-11 — [18F]PSMA-11 PET/CT
Diagnostic Test: [68Ga]PSMA-11 — [68Ga]PSMA-11 PET/CT

SUMMARY:
Prostate cancer (PCa) is the most frequently occurring male cancer in Belgium. After treatment with surgery and/or radiotherapy, almost half of the patients suffer from a tumor recurrence, often diagnosed by an increase in serum tumor marker Prostate Specific Antigen (PSA) within the first few years after primary treatment. However, for salvage therapy to be successful, precise localization of metastases is necessary to determine the most appropriate treatment. In so-called oligo-metastatic disease targeted therapy may still be curative and prevent the disease from spreading to distant locations. Therefore it is of paramount importance to have an accurate tool of medical imaging to localize all possible locations to be treated.

Recently, prostate specific membrane antigen (PSMA) has gained interest for PCa-specific imaging. Due to overexpression of PSMA in both primary and metastatic PCa, radiotracers targeting this protein have shown an increased selectivity and sensitivity compared to conventional imaging. The main objective of this phase 3 trial is to determine the position of [18F]PSMA-11 PET/CT within the field of available radiotracers for diagnosis of prostate cancer. For this, the diagnostic performances of [18F]PSMA-11 will be compared to those of the current state-of-the-art radiotracer [68Ga]PSMA-11.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with prostate cancer, either in the setting of diagnosis of biochemical recurrence after previous treatment, or at primary diagnosis and staging.

Exclusion Criteria:

* Age < 18 years
* Physically or mentally unfit to perform the sequential procedures
* Refusal of patient to be informed about accidental findings on scans
* History of anaphylactic shock after administration of Visipaque CT contrast
* Serum creatinine concentration > 2.0 mg/dl and/or estimated glomerular filtration rate < 60 ml/min.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male with prostate cancer
Enrollment: 96 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the non-inferiority of [18F]PSMA-11 compared to [68Ga]PSMA-11 with respect to the number of positive PET scans. Hereby, a positive PET scan is defined as a scan showing at least one suspected lesion. | 0 to 100 minutes post injection for both [18F]PSMA-11 and [68Ga]PSMA-11
  The non-inferiority of [18F]PSMA-11 will be investigated based on a Tango's score two-sided 95% confidence interval (CI) for a difference of proportions of positive scans of [18F]PSMA-11 compared to [68Ga]PSMA-11 with matched pairs. Non-inferiority will be concluded if the lower limit of this CI is larger than 0.10 (non-inferiority limit).

SECONDARY OUTCOMES:
Evaluation of the superiority of [18F]PSMA-11 compared to [68Ga]PSMA-11 with respect to the number of positive PET scans. Hereby, a positive PET scan is defined as a scan showing at least one suspected lesion. | 0 to 100 minutes post injection for both [18F]PSMA-11 and [68Ga]PSMA-11
  Superiority of [18F]PSMA-11 compared to [68Ga]PSMA-11 with respect to the number of positive PET scans will be statistically assessed by applying a McNemar's test on the proportions of positive PET scans in each group. Hereby, superiority is defined as a difference of minimum 10% in the proportions of positive PET scans ([18F]PSMA-11 > [68Ga]PSMA-11).
Evaluation of the superiority of [18F]PSMA-11 compared to [68Ga]PSMA-11 with respect to the total number of suspected prostate cancer lesions in corresponding ([68Ga]PSMA-11 vs [18F]PSMA-11) scans. | 0 to 100 minutes post injection for both [18F]PSMA-11 and [68Ga]PSMA-11
  The McNemar-Bowker test of symmetry of k X k contingency tables will be applied to investigate differences between [18F]PSMA-11 and [68Ga]PSMA-11 scans. Hereby, the superiority is defined as a difference of minimum 10% ([18F]PSMA-11 > [68Ga]PSMA-11).
Evaluation of the superiority of [18F]PSMA-11 compared to [68Ga]PSMA-11 with respect to the scoring of corresponding ([68Ga]PSMA-11 vs [18F]PSMA-11) suspected lesions. | 0 to 100 minutes post injection for both [18F]PSMA-11 and [68Ga]PSMA-11
  The McNemar-Bowker test of symmetry of k X k contingency tables will be applied to investigate differences between [18F]PSMA-11 and [68Ga]PSMA-11 scans. Hereby, the superiority is defined as a difference of minimum 10% ([18F]PSMA-11 > [68Ga]PSMA-11).
Descriptive evaluation of [18F]PSMA-11 compared to [68Ga]PSMA | 0 to 100 minutes post injection for both [18F]PSMA-11 and [68Ga]PSMA-11
  This endpoint will be examined in the total group of patients, as well as in a subgroup of patients with a specific disease stage including primary diagnosis, castrate sensitive biochemical recurrence, and castrate resistant biochemical recurrence. Additionally, within these subgroups, a further subdivision can be made on the basis of a specific location of the suspected lesions, PSA values, PSA doubling times and metastatic disease burden).
Evaluation of the diagnostic specificity of [18F]PSMA-11 compared to [68Ga]PSMA-11 | 0 to 180 days post [18F]PSMA-11 and [68Ga]PSMA-11 administration
  This endpoint will be evaluated in a descriptive way, more specifically by a description of the number of positive scans (and/or positive lesions) that can be confirmed via an anatomopathological diagnosis, changes in PSA concentration or via MRI, and by comparison of these numbers between [18F]PSMA-11 and [68Ga]PSMA-11.
Evaluation of the safety of [18F]PSMA-11 administration: CTCAE 4.0 criteria | 0 to 24 h post [18F]PSMA-11 and [68Ga]PSMA-11 administration
  Adverse events will be reported and scored (CTCAE 4.0 criteria) between the first dose administration of trial medication and the last trial related activity. From the time of radiotracer injection till completion of the PET/CT scan (for both [18F]PSMA-11 and [68Ga]PSMA-11), the site staff will visually observe and actively ask the patient whether or not he has observed any adverse effects. Although [18F]PSMA-11 is totally eliminated from the body within 9 hours post injection (= 10 x half-life of 47 ± 5 minutes), AE's occurring up to 24h after the second PET/CT scan will also be handled as such if spontaneously reported by the patient to the investigator.
Assessment of the interobserver variability with regard to the evaluation of the [18F]PSMA-11 and [68Ga]PSMA-11 PET scans | 0 to 100 minutes post injection for both [18F]PSMA-11 and [68Ga]PSMA-11
  This endpoint will be evaluated by determining a Cohen's kappa value

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, Prof., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium